CLINICAL TRIAL: NCT03555448
Title: Once a Day Immunosuppression Regimen: Outcomes and Compliance
Brief Title: Once Daily Immunosuppression Regimen
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: poor recruitment during pandemic and after
Sponsor: Washington University School of Medicine (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201803162
Record Dates: First submitted 2018-05-17; First posted 2018-06-13 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Kidney Transplant; Complications
Keywords: Immunosuppression

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Once daily regimen (Active Comparator): Once daily medication regimen (Envarsus and azathioprine)
  Interventions: Drug: Once daily immunosuppression regimen
- Twice daily regimen (Active Comparator): Twice daily medication regimen (Tacrolimus and mycophenolic acid)
  Interventions: Drug: Twice daily immunosuppression regimen

INTERVENTIONS:
Drug: Once daily immunosuppression regimen — Intervention focuses on the type of regimen, in this case the intervention arm will receive a once daily regimen for immunosuppression compared to the twice daily regimen.
  Arms: Once daily regimen
Drug: Twice daily immunosuppression regimen — This is the arm which we are designating the standard, which will be the comparison to the active drug arm.
  Arms: Twice daily regimen

SUMMARY:
The purpose of this research study is to determine whether an immunosuppressive maintenance regimen of Envarsus/azathioprine compared to a tacrolimus/ mycophenolic acid regimen is associated with better compliance, tolerability, and lower biopsy proven rejection.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years old
* Kidney transplant recipient
* Thymoglobulin induction

Exclusion Criteria:

* Non-renal organ transplant
* Combined organ transplant
* Inability to receive Envarsus after transplant
* Discharged to acute care facility after transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rowena Delos Santos, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Budde K, Bunnapradist S, Grinyo JM, Ciechanowski K, Denny JE, Silva HT, Rostaing L; Envarsus study group. Novel once-daily extended-release tacrolimus (LCPT) versus twice-daily tacrolimus in de novo kidney transplants: one-year results of Phase III, double-blind, randomized trial. Am J Transplant. 2014 Dec;14(12):2796-806. doi: 10.1111/ajt.12955. Epub 2014 Oct 2. PMID 25278376
- [Background] Bunnapradist S, Ciechanowski K, West-Thielke P, Mulgaonkar S, Rostaing L, Vasudev B, Budde K; MELT investigators. Conversion from twice-daily tacrolimus to once-daily extended release tacrolimus (LCPT): the phase III randomized MELT trial. Am J Transplant. 2013 Mar;13(3):760-9. doi: 10.1111/ajt.12035. Epub 2012 Dec 21. PMID 23279614
- [Background] Jamieson NJ, Hanson CS, Josephson MA, Gordon EJ, Craig JC, Halleck F, Budde K, Tong A. Motivations, Challenges, and Attitudes to Self-management in Kidney Transplant Recipients: A Systematic Review of Qualitative Studies. Am J Kidney Dis. 2016 Mar;67(3):461-78. doi: 10.1053/j.ajkd.2015.07.030. Epub 2015 Sep 11. PMID 26372087
- [Background] Laliberte F, Nelson WW, Lefebvre P, Schein JR, Rondeau-Leclaire J, Duh MS. Impact of daily dosing frequency on adherence to chronic medications among nonvalvular atrial fibrillation patients. Adv Ther. 2012 Aug;29(8):675-90. doi: 10.1007/s12325-012-0040-x. Epub 2012 Aug 15. PMID 22898791
- [Background] Rostaing L, Bunnapradist S, Grinyo JM, Ciechanowski K, Denny JE, Silva HT Jr, Budde K; Envarsus Study Group. Novel Once-Daily Extended-Release Tacrolimus Versus Twice-Daily Tacrolimus in De Novo Kidney Transplant Recipients: Two-Year Results of Phase 3, Double-Blind, Randomized Trial. Am J Kidney Dis. 2016 Apr;67(4):648-59. doi: 10.1053/j.ajkd.2015.10.024. Epub 2015 Dec 22. PMID 26717860
- [Background] Vrijens B, Heidbuchel H. Non-vitamin K antagonist oral anticoagulants: considerations on once- vs. twice-daily regimens and their potential impact on medication adherence. Europace. 2015 Apr;17(4):514-23. doi: 10.1093/europace/euu311. Epub 2015 Feb 17. PMID 25694538

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Once Daily Regimen | Twice Daily Regimen
Started | 25 | 26
Completed | 23 | 24
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Once Daily Regimen | Twice Daily Regimen | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.58 (12.3) | 55.6 (14.3) | 56.55 (12.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 11 | 15 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 4 | 12
  White | 15 | 19 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Change in Compliance and Tolerability of Medication Regimen at 3 and 12 Months
Description: BAASIS Survey
Time Frame: 3 months and 12 months post transplant
Measure: Number; unit: participants
Arm/Group | Once Daily Regimen | Twice Daily Regimen
Number analyzed (Participants) | 23 | 24
participants
  3month:Q1 Do you recall not having taken your immunosuppressive meds some times in the past 4 weeks? | 1 | 2
  3month:Q2 Have you skipped several consecutive doses of immunosuppressive meds in the past 4 weeks? | 0 | 0
  3month:Q3 Do you recall taking immunos meds with >2hrs from the prescribed time in the past 4 weeks? | 9 | 5
  3month:Q4 Have you reduced the prescribed amount of immunosuppressive meds during the past 4 weeks? | 1 | 0
  12month:Q1 Do you recall not having taken your immunosuppressive meds some times in past 4 weeks? | 1 | 2
  12month:Q2 Have you skipped several consecutive doses of immunosuppressive meds in the past 4 weeks? | 0 | 1
  12mth:Q3 Do you recall taking immunos meds with >2hrs from the prescribed time in the past 4 weeks? | 3 | 6
  12month:Q4 Have you reduced the prescribed amount of immunosuppressive meds during the past 4 weeks? | 0 | 0

2. Secondary Outcome: Change in Self-recorded Compliance and Tolerability of Medication Regimen at 3 and 12 Months
Description: Pill Manager (personal medication record keeping for those who participants who choose to use this method of recording their self-administered medication)
Time Frame: 3 months and 12 months post transplant
Population: There are Zero "0" patients in study who used the pill manager during the study. No data were collected
Arm/Group | Once Daily Regimen | Twice Daily Regimen
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Composite Endpoint Measurement
Description: Number of Participants with Biopsy proven Acute Rejection, graft loss, death, Lost to follow-up at 12 months.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Once Daily Regimen | Twice Daily Regimen
Number analyzed (Participants) | 23 | 24
participants | 1 | 1

ADVERSE EVENTS:
Time Frame: 1 year from time of transplant
Arm/Group | Once Daily Regimen | Twice Daily Regimen
All-Cause Mortality (participants affected / at risk) | 1/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 9/23 | 13/24
Other Adverse Events (participants affected / at risk) | 1/23 | 1/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Once Daily Regimen (N=23) | Twice Daily Regimen (N=24)
AKI (Renal and urinary disorders) | 2 (3) | 3 (3)
Infection (Infections and infestations) | 3 (4) | 3 (3)
Urine leak (Renal and urinary disorders) | 0 (0) | 1 (1)
Hyperkalemia (General disorders) | 1 (1) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nausea and vomiting/abdominal pain (Gastrointestinal disorders) | 4 (5) | 3 (3)
Transplant renal artery stenosis (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Once Daily Regimen (N=23) | Twice Daily Regimen (N=24)
Dialysis access issue (clotting/bleeding) (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT03555448/Prot_SAP_000.pdf